CLINICAL TRIAL: NCT00824759
Title: Cardioprotective Effects of Increased Endogenous Erythropoietin After Normobaric Oxygen Breathing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because it seemed not of interest based on the current literature
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Momeni, MD; Chef de Clinique Adjointe, Department of Anesthesiology, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/24NOV/331
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Healthy; Coronary Artery Bypass Graft
Keywords: Healthy subjects; CABG; Patients undergoing coronary artery bypass graft under cardiopulmonary bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Other: pure oxygen breathing versus air
- oxygen (Active Comparator)
  Interventions: Other: pure oxygen breathing versus air

INTERVENTIONS:
Other: pure oxygen breathing versus air — one group will breath pure oxygen; the other will breath air

SUMMARY:
Tissue hypoxia is the only accepted trigger for erythropoietin (EPO) production. However, in healthy subjects EPO concentrations have also increased after oxygen breathing. The aim of our study is to confirm these observations.

Besides its main function in erythropoiesis, EPO has also shown tissue protective effects. The second goal of our study is to observe the cardioprotective effects of increased endogenous EPO, induced after normobaric oxygen breathing.

DETAILED DESCRIPTION:
Currently, renal tissue hypoxia is the only widely accepted trigger for erythropoietin (EPO) production. However, previous studies in healthy subjects have demonstrated that a sudden and sustained decrease in tissue oxygen level, aside from an absolute low level of tissue oxygen tension, could also act as a trigger for EPO production. To confirm these observations and to clarify an eventual role of free oxygen radicals and antioxidants, hypobaric pure oxygen will be administered to healthy subjects.

The major physiologic function of EPO is thought to be the induction of erythropoiesis. However, a growing body of evidence indicates that EPO has tissue-protective effects and prevents tissue damage during ischemia. In an ex vivo proof-of-concept, protective effects of EPO have been shown in human myocardium.

The second goal of our study is to observe the cardioprotective effects of increased endogenous EPO, induced after normobaric oxygen breathing.

ELIGIBILITY:
Inclusion Criteria:

* healthy non-smokers; patients undergoing CABG under cardiopulmonary bypass

Exclusion Criteria:

* Subjects with a pulmonary disease; subjects who have stayed at high altitude since at least 3 months; healthy subjects taking medication; patients undergoing a redo or combined cardiac surgery; patients with renal insufficiency; any emergency CABG; Patients with pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
decrease in Troponin-I values | 12h

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Background] Balestra C, Germonpre P, Poortmans JR, Marroni A. Serum erythropoietin levels in healthy humans after a short period of normobaric and hyperbaric oxygen breathing: the "normobaric oxygen paradox". J Appl Physiol (1985). 2006 Feb;100(2):512-8. doi: 10.1152/japplphysiol.00964.2005. Epub 2005 Oct 20. PMID 16239610
- [Background] Parsa CJ, Matsumoto A, Kim J, Riel RU, Pascal LS, Walton GB, Thompson RB, Petrofski JA, Annex BH, Stamler JS, Koch WJ. A novel protective effect of erythropoietin in the infarcted heart. J Clin Invest. 2003 Oct;112(7):999-1007. doi: 10.1172/JCI18200. PMID 14523037